CLINICAL TRIAL: NCT01813656
Title: A Multiple-Center, Randomized, Double-Blind Study of Aripiprazole for Treatment of Methamphetamine Dependence
Brief Title: An Study of Aripiprazole in the Treatment of Methamphetamine Dependence
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Aripiprazole arm had obvious adverse reactions,especially akathisia.
Sponsor: Wei Hao (Other)
Responsible Party: Sponsor-Investigator, Wei Hao, The Second Xiangya Hospital of Cental South University, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100000-068942
Record Dates: First submitted 2012-11-28; First posted 2013-03-19 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Methamphetamine Dependence
Keywords: Methamphetamine-Associated Psychosis; Aripiprazole
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Experimental): Aripiprazole arm,5mg/pill,10mg/day.last12weeks.
  Interventions: Drug: Aripiprazole
- Sugar pill (Placebo Comparator): placebo arm,5mg/pill,10mg/day,last12weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole group,5mg/pill,10mg/day non-forced titration method,last 12weeks
  Other Names: Aopai H20041507
  Arms: Aripiprazole
Drug: placebo — placebo group,5mg/pill,10mg/day non-forced titration method,last 12 weeks
  Arms: Sugar pill

SUMMARY:
Methamphetamine substance use is common worldwide. No approved pharmacologic treatments for methamphetamine dependence exist. Aripiprazole are Second generation antipsychotics，but have different pharmacological effects of neurotransmitters.To determine whether mirtazapine would reduce methamphetamine use among mehtamphetamine addicts.

DETAILED DESCRIPTION:
Methods:A Multiple-Center, Randomized, Double-Blind.

ELIGIBILITY:
Inclusion Criteria:

1. Patients,Diagnostic and Statistical Manual of Mental Disorders 4thed. (DSM-IV) criteria for Methamphetamine dependence.
2. Must sign a Information consent form.
3. Required to provide detailed address and phone number

Exclusion Criteria:

1. Serious organic disease.
2. Suicide ideation or hurt others.
3. Taking antipsychotic within two weeks before.
4. drug allergy to Risperidone or Aripiprazole.
5. pregnancy and breastfeeding women.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
abstinent time of Methamphetamine addict | up to 3 months
  methamphetamine-positive urine test results,self-reports of substance use

SECONDARY OUTCOMES:
number of Participants with Adverse Events as a Measure of Safety and Tolerability | up to 3 months
  use Abnormal Involuntary Movement Scale ,Simpson-Angus Scale and Barnes akathisia Scale

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hao, MD., Ph.D., Study Director — Central South University
Locations (1):
- The Second Xiangya Hospital of Central University, Changsha, Hunan, China